CLINICAL TRIAL: NCT06313021
Title: Examination of the Validity and Reliability of the Turkish Version of the Brief Assessment of Cognitive Impairment in Individuals With Stroke Scale
Brief Title: Turkish Version of the Brief Assessment of Cognitive Impairment in Individuals With Stroke Scale
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Birol Onal, Assistant professor, Ataturk University
Other Study IDs: 2023.12.03
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Cognition
Keywords: stroke; cognition; validity; reliability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke group: stroke group
  Interventions: Other: Reliability and Validity Study

INTERVENTIONS:
Other: Reliability and Validity Study — Reliability and Validity Study

SUMMARY:
Cognitive processing involves many interrelated cognitive domains, such as performing daily tasks, attention, language, and memory. 70% of individuals with stroke experience cognitive problems. Due to cognitive problems, individuals with stroke have difficulty processing and planning information. This situation negatively affects daily living activities and returning to work. Cognitive disorders that occur after stroke negatively affect the functional independence of individuals. At the same time, individuals with stroke have difficulty structuring and organizing information. The individual may not be able to pay sufficient attention during the activity in terms of planning, automatic attention and adaptation to the stages required by the job.

Cognitive evaluation should include cognition, orientation, and higher cortical functions because the cognitive process is a very complex process. Assessment methods frequently used in cognitive evaluation of stroke patients; Scales and tests such as Simple Mental Test, Mini Mental State Test, Montreal Cognitive Assessment Scale, Wechsler Memory and Intelligence Test are used. General problems with these evaluations; Some of them have a long application period, some of them have problems in perception of the patients, and some of them have a low power to distinguish the cognitive problems of the patients. When the Brief Assessment of Cognitive Impairment Scale, a newly introduced scale in the literature, is examined; It attracts attention because the items are very simple for patients to perceive, combine cognitive tests and cognitive questionnaires, have a short application period, and have not shown a ceiling or floor effect in previous studies. For all these reasons, this study was planned to conduct the Turkish validity and reliability study of the Brief Assessment of Cognitive Impairment Scale.

DETAILED DESCRIPTION:
Cognition; It is a broad concept that includes mental processes such as an individual's perception, understanding, processing and remembering of information. Cognition includes many mental activities such as thinking, learning, memory, problem solving, attention, and language use. The importance of cognition is related to the individual's ability to understand his environment, learn, solve problems and make effective decisions in daily life. These processes can have a direct impact on an individual's education, work, relationships, and overall quality of life. Therefore, understanding and supporting cognition can help individuals manage and improve their lives more effectively.

A common consequence of stroke is impaired cognition. It is stated that in the three-year period after stroke, up to 39% of patients have cognitive impairment. There is a significant relationship between cognitive abilities and functional performance. Therefore, cognitive impairment may reduce the independence of people with stroke in performing basic activities of daily living (such as eating, dressing, and toileting) and activities of daily living (such as household chores and social interactions). As a result, people with post-stroke cognitive impairment often require ongoing care and support, which can put pressure on caregivers and society. Therefore, effective assessment of post-stroke cognition is crucial for stroke rehabilitation. Frequently used assessment methods in the cognitive evaluation of stroke patients include scales and tests such as Mini Mental State Test, Montreal Cognitive Assessment Scale, and Wechsler Memory and Intelligence Test. However, when these evaluations are examined, there are problems in detecting the cognitive effects of patients with different severities due to the long application times of some of them and the floor and ceiling effects in some of them. Therefore, we planned this study to test the Turkish validity and reliability of the Brief Assessment of Cognitive Impairment Scale, a new, simple diagnostic tool that combines cognitive tests and cognitive questionnaires, in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 40 and 75,
* Individuals who volunteer to participate in the research,
* Individuals diagnosed with stroke,
* Individuals who do not have cooperation and communication problems

Exclusion Criteria:

* Those with neurological problems other than stroke (patients diagnosed with Alzheimer's, Parkinson's, Dementia, MS)
* Those with perceptual problems
* Individuals with cooperation and communication problems

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will consist of individuals with stroke over the age of 40 who come to the University Hospital for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Brief Assessment of Cognitive Impairment Scale | seven day
  The Brief Assessment of Cognitive Impairment was developed by Danish researchers to assess cognitive impairment and dementia. To practice BASIC, one needs a registration form, a picture card, a manual, and a stopwatch, like the stopwatch in our smartphone's clock app. BASIC consists of five parts: presentation of pictures for memory testing, patient-directed questions, fluency in naming supermarket products, recall of pictures, and assessor-directed questions. Assessor-directed questions can be administered before, during, or after the patient is evaluated. It is performed for evaluation in an environment free from distractions and with adequate lighting. If the patient uses glasses or hearing aids, these must be present. It is necessary to explain the purpose of the evaluation to the patient. The test consists of 11 questions. The lowest score is 0, the highest score is 25. As the score decreases, cognitive status worsens.

SECONDARY OUTCOMES:
Mini Mental State Test | seven day
  The test develoThe test developed by Folstein et al. in 1975 is the most widely used cognitive screening test. The test consists of 11 items; It is evaluated out of 30 points: 10 points for time and space orientation, 6 points for memory, 5 points for attention, 8 points for language and 1 point for visual-spatial function. 24-30 points are considered normal, 18-23 points are considered mild cognitive impairment, 12-17 points are considered moderately severe, and below 12 points are considered severe cognitive impairment. A standardized MMDT was created for the Turkish society and validity and reliability tests were conducted.
Sociodemographic Assessment | seven day
  Before individuals; Parameters such as age, gender, marital status, educational status, profession, Brunnstrom level, stroke duration, side of stroke, affected vein, dominant extremity, smoking and alcohol use, assistive devices used, CV information, family history information and medications used will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Birol Önal, Dr, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)